CLINICAL TRIAL: NCT06282939
Title: Optima Coil Performance in The Interventional Management of Intracranial Aneurysms Registry
Acronym: OPTIMA
Status: Recruiting | Type: Observational
Sponsor: HCA Healthcare Research Institute (Other)
Collaborators: Balt USA (Industry)
Responsible Party: Sponsor
Other Study IDs: 20234314
Record Dates: First submitted 2023-11-06; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: OPTIMA and OPTIMAX Coils manufactured by Balt USA — *Percentage from protocol

SUMMARY:
This is a prospective, open-label, consecutive enrollment, multi-center, U.S. registry of patients with intracranial aneurysms who are treated with the Optima Coil System.

The primary objective of this registry is to evaluate the safety and effectiveness of the OptimaTM Coil System, including the OptiMAX Coils, in the real-world treatment of intracranial aneurysms. Imaging will be analyzed by a designated core neuroimaging lab to assess procedural success and aneurysm occlusion rates. Intent to treat population total: 700 patients 600 patients, up to 100 screen failures.

DETAILED DESCRIPTION:
The primary objective of this registry is to evaluate the safety and effectiveness of the OptimaTM Coil System, including the OptiMAX Coils, in the real-world treatment of intracranial aneurysms. Imaging will be analyzed by a designated core neuroimaging lab to assess procedural success and aneurysm occlusion rates.

The core lab will consist of 4-5 physicians, 2-3 from within HCA Healthcare, and 2-3 from outside of HCA Healthcare. Core lab physicians will be blinded to patient characteristics for HIPAA compliance. Physicians within the core lab will not be principal investigators enrolling patients in the study.

600 subjects with intracranial saccular aneurysms (maximum dimension ≤ 24 mm), ruptured or unruptured, treated with the OptimaTM Coil System.

As this is a registry, there will be no formal hypothesis testing of the study endpoints, and no formal sample size / power calculations will be performed.

Approximately 600 subjects will be enrolled in the registry at up to 12 clinical sites in the US. Data analyses will be performed and led by the study PIs, Site PIs, and Sub-investigators.

Expected descriptive statistics will include baseline patient demographics, procedural characteristics, radiographic parameters, safety outcomes, clinical and efficacy outcomes. Pilot univariate and multivariate logistic regression will be performed on the intention-to-treat cohort to identify predictors of adequate and complete aneurysm occlusion.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in this registry must be treated in accordance with the FDA-cleared indication for the Optima Coil System.

In addition:

1. Patient age ≥ 18 years;
2. Candidate aneurysm is a previously untreated, saccular intracranial aneurysm measuring ≤ 24 mm in maximal diameter and suitable for embolization with coils;
3. OptimaTM coil system accounts for at least 75% of the total number of implanted coils;
4. Patient/ LARreceived the IRB-approved Consent Information Sheet to augment clinical procedure consent, and provided verbal consent to participate in the study
5. Subject willing to comply with the protocol follow-up requirements; and
6. Hunt & Hess classification of equal to or less than 4 for ruptured aneurysms, if applicable.

Exclusion Criteria:

Since this is a real-world registry, few exclusion criteria are defined. Adjustments for baseline patient characteristics and aneurysm morphology will be used to identify outliers and unique cohorts.

1. Life expectancy less than 1 year.
2. Patient previously enrolled in the OPTIMA Registry.
3. Known multiple intracranial aneurysms, apart from the targeted aneurysm for the OPTIMA study, requiring treatment during the index procedure or within the study follow-up period.
4. Patient is unwilling or unable to comply with the protocol follow-up schedule and/or based on the Investigator's judgment the patient is not a good registry candidate.
5. Participation in another confirmed interventional clinical study that could confound the evaluation of this registry, per PI discretion.
6. Pre-planned staged procedures on unruptured target aneurysms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 600 subjects with intracranial saccular aneurysms (maximum dimension ≤ 24 mm), ruptured or unruptured, treated with the OptimaTM Coil System.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Measure Adequate Occlusion Using modified Raymond-Roy Occlusion Class (MRRC) I and II score | 1 year follow up +/- 90 days
  Rated by a designated core lab without retreatment as confirmed by core lab adjudication.
Assess coiling alone or in combination with adjunctive devices for approximately 400 patients | 1 year follow up +/- 90 days
  Subgroup using adjunctive devices include including balloon remodeling and stenting
Evaluate Coiling with flow diversion for approximately 200 subjects | 1 year follow up +/- 90 days
  Subgroup utilizing flow diverter for approximately 200 subjects
Subgroup analyses will be performed examining: | 1 year follow up +/- 90 days
  Aneurysms treated predominantly (≥50%) with Balt manufactured coils will also be analyzed for the number of coils utilized per aneurysm and procedure duration
Analyze outcomes of small aneurysms defined as smaller than 5mm | 1 year follow up +/- 90 days
  Outcomes of small aneurysms defined as smaller than 5mm

SECONDARY OUTCOMES:
Adequate occlusion | Immediate Post Procedure
  Confirmed by core lab adjudication.
Packing density | Day 1
  The percentage of coil volume to aneurysm volume using AngioSuite.
Complete occlusion | 1 Year post- procedure
  Utilizing MRRC Class I
Complete occlusion | Immediate post procedure
  Utilizing MRRC Class 1
Recanalization rate | 1 year post procedure
  Any worsening in aneurysm occlusion on the MRRC scale
Retreatment rate | 1 year post procedure
  Retreatment of Target aneurysm
Change in degree of disability | 1 year post procedure
  The proportion of patients with modified Rankin Scale score 0-2 (or at baseline score if >2)
The number of coils used in an aneurysm | Upon enrollment
  The number of coils used in an aneurysm stratified by aneurysm size.
Procedural fluoroscopic time | During procedure
  Procedural fluoroscopic time

OTHER OUTCOMES:
Primary Safety Endpoint | 7 days post-procedure or discharge
  Device-related SAE
Secondary Safety Endpoint | 12 months post enrollment
  1. Intraprocedural aneurysm perforation or rupture.
  2. Intraprocedural symptomatic thromboembolic event.
  3. All-cause mortality at 12 months post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yoo, Principal Investigator — HCA Research Institute
Locations (1):
- Med City Plano, Plano, Texas, United States